CLINICAL TRIAL: NCT02390063
Title: A Randomized Phase I Study to Determine the Safety and Immunogenicity of ChAd-MVA Vaccination Compared to MVA Alone With and Without Low Dose Cyclophosphamide in Low and Intermediate Risk Localised Prostate Cancer
Brief Title: Vaccination in Prostate Cancer (VANCE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: VANCE01
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — TroVax; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- CHAMVA standard regime (Experimental): ChAdOx1.5T4 prime followed by two boost of MVA.5T4 vaccine at 4 week intervals until radical prostatectomy
  Interventions: Biological: ChAdOx1.5T4; Biological: MVA.5T4
- CHAMVA+CTX standard regime (Experimental): One week of low dose cyclophosphamide pre-conditioning before each vaccination. ChAdOx1.5T4 prime followed by two boost of MVA.5T4 at 4 week intervals until radical prostatectomy.
  Interventions: Biological: ChAdOx1.5T4; Biological: MVA.5T4; Drug: Cyclophosphamide
- MVA standard regime (Active Comparator): Three MVA.5T4 vaccinations at 4 week intervals until radical prostatectomy
  Interventions: Biological: MVA.5T4
- MVA+CTX standard regime (Active Comparator): One week of low dose cyclophosphamide pre-conditioning before each vaccination.Three MVA.5T4 vaccinations at 4 week intervals until radical prostatectomy
  Interventions: Biological: MVA.5T4; Drug: Cyclophosphamide
- CHAMVA accelerated regime (Experimental): ChAdOx1.5T4 prime followed by one boost of MVA.5T4 one week later until radical prostatectomy.
  Interventions: Biological: ChAdOx1.5T4; Biological: MVA.5T4
- CHAMVA+CTX accelerated regime (Experimental): One week of low dose cyclophosphamide pre-conditioning before each vaccination. ChAdOx1.5T4 prime followed by one boost of MVA.5T4 one week later until radical prostatectomy.
  Interventions: Biological: ChAdOx1.5T4; Biological: MVA.5T4; Drug: Cyclophosphamide
- CHAMVA accelerated regime AS (Experimental): ChAdOx1.5T4 prime followed by one boost of MVA.5T4 one week later. Patients continue on active surveillance.
  Interventions: Biological: ChAdOx1.5T4; Biological: MVA.5T4
- CHAMVA+CTX accelerated regime AS (Experimental): One week of low dose cyclophosphamide pre-conditioning before each vaccination. ChAdOx1.5T4 prime followed by one boost of MVA.5T4 one week later. Patients continue on active surveillance.
  Interventions: Biological: ChAdOx1.5T4; Biological: MVA.5T4; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: ChAdOx1.5T4 — A recombinant simian adenovirus encoding human tumour-associated antigen 5T4
  Arms: CHAMVA accelerated regime; CHAMVA accelerated regime AS; CHAMVA standard regime; CHAMVA+CTX accelerated regime; CHAMVA+CTX accelerated regime AS; CHAMVA+CTX standard regime
Biological: MVA.5T4 — A recombinant replication deficient Modified Vaccinia Ankara virus encoding human tumour-associated antigen 5T4
Drug: Cyclophosphamide — Metronomic cyclophosphamide (50mg bd)
  Other Names: CTX, CY, Cytoxan
  Arms: CHAMVA+CTX accelerated regime; CHAMVA+CTX accelerated regime AS; CHAMVA+CTX standard regime; MVA+CTX standard regime

SUMMARY:
This is a clinical trial of a new treatment for prostate cancer that is a type of vaccine that could be a new way to treat cancer. A vaccine that could alert the immune system to the presence of cancer cells in the body may enable the immune system to target and kill those cells effectively. This vaccine is intended to work by making the immune system kill cells that have a special protein (called 5T4) that is present on the surface of cancer cells. The vaccine is made up of two recombinant viruses ("ChAdOx1" and "MVA") that have been designed to produce the 5T4 protein and have been modified so that they are weakened and cannot reproduce themselves within the body like normal viruses. Once injected into the body, these viruses make the 5T4 protein and help the body's immune system to learn to target this protein and destroy cancer cells.

This is a first-in-human study to evaluate the safety and immunogenicity of ChAdOx1.5T4-MVA.5T4 vaccination regime. It is evaluated in neo-adjuvant setting in low and intermediate risk localised prostate cancer patients who have either decided to have their prostate removed or are stable on active surveillance.

ELIGIBILITY:
Inclusion Criteria(Radical Prostatectomy patients):

* Males aged 18 years and older
* Histologically confirmed prostate cancer diagnosed on biopsy within 6 months
* Clinically localised, low or intermediate risk prostate cancer, i.e.:

  * Gleason score ≤ 7
  * Local tumour stage ≤T2c
  * No evidence of metastases (Nx/N0 and Mx/M0)
  * PSA ≤ 20 ng/ml
* Scheduled for and considered fit for radical prostatectomy
* Absence of any indication to perform urgent surgery that would not allow administration of the vaccine during the 12 week period prior to radical prostatectomy
* No invasive treatment for prostatic disease within the last 2 years
* Subject is free of clinically apparent/active autoimmune disease (no prior confirmed diagnosis or treatment for autoimmune disease including Systemic Lupus Erythematosis, Grave's Disease, Hashimoto's Thyroiditis, Multiple Sclerosis, and Insulin Dependent Diabetes Mellitus). Note subjects with Non-Insulin Dependent Diabetes Mellitus can be included.
* Subject has adequate bone marrow function as defined by an Absolute Lymphocyte Count (ALC) ≥ 500/µL, Absolute Neutrophil Count (ANC) >1200/µL, Platelet Count >100,000/µL.
* Subject must practice a reliable form of contraception (barrier or vasectomy) while they are being treated with vaccines and another effective method of birth control must also be used by their partner

Inclusion Criteria (Active Surveillance patients)

* Males aged 18 and older
* Histologically confirmed prostate cancer diagnosed on biopsy within 6 months
* Clinically localised, low or intermediate risk prostate cancer, i.e.:

  * Gleason score ≤ 7
  * Local tumour stage ≤T2c
  * No evidence of metastases (Nx/N0 and Mx/M0)
  * PSA ≤ 20 ng/ml
* Stable disease on Active Surveillance for a minimum of 12 months previously
* Suitable to remain on Active Surveillance at time of last clinical assessment
* No invasive treatment for prostatic disease within the last 2 years
* Subject is free of clinically apparent/active autoimmune disease (no prior confirmed diagnosis or treatment for autoimmune disease including Systemic Lupus Erythematosis, Grave's Disease, Hashimoto's Thyroiditis, Multiple Sclerosis, and Insulin Dependent Diabetes Mellitus). Note subjects with Non-Insulin Dependent Diabetes Mellitus can be included.
* Subject has adequate bone marrow function as defined by an Absolute Lymphocyte Count (ALC) ≥ 500/µL, Absolute Neutrophil Count (ANC) >1200/µL, Platelet Count >100,000/µL.
* Subject must practice a reliable form of contraception (barrier or vasectomy) while they are being treated with vaccines and another effective method of birth control must also be used by their partner

Exclusion Criteria:

* Diagnosis of any cancer other than prostate cancer within the last 5 years (except basal cell carcinoma)
* Any suspicion of metastatic cancer
* Any Gleason grade 5 component in the prostatic biopsies
* Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Seropositive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) or HIV
* Any confirmed or suspected immunosuppressive or immunodeficient state, asplenia, recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled/topical steroids are allowed)
* Platelet count >400,000/μL; Monocytes >80,000/μL; Hemoglobin <11g/dL
* Known allergy to neomycin
* History of allergic response to previous vaccinia vaccinations
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products
* History of hypersensitivity and haemorrhagic cystitis
* Any history of anaphylaxis
* Suspected or known current injecting drug or alcohol abuse (as defined by an alcohol intake of greater than 42 units per week)
* History of a serious psychiatric condition or other circumstance s that may be associated with not understanding or complying with the study protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2018-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Vaccine safety and immunogenicity | Up to 52 weeks
  Development or increase in anti-5T4 cellular and humoral responses in patients treated with CHAMVA or CHAMVA + CTX

SECONDARY OUTCOMES:
Cellular and humoral immune response with CHAMVA | Up to 52 weeks
  Development or increase in anti-5T4 cellular and humoral responses in patients treated with the CHAMVA vaccination regimes
Cellular and humoral immune response with MVA | Up to 52 weeks
  Development or increase in anti-5T4 cellular and humoral response in patients treated with the MVA vaccination regimes.
PSA level change secondary to vaccination | Participants will be followed for the duration of the study, up to 52 weeks
  PSA level decrease in patients treated with CHAMVA or MVA vaccination at week 4,8 or 12.
MRI or Gleason score change secondary to vaccination | Participants will be followed for the duration of the study, up to 52 weeks
  Reduction of tumour burden or Gleason score at weeks 4, 8 or 12.
Regulatory T-cell response | Participants will be followed for the duration of the study, up to 52 weeks
  Change in the frequency of regulatory T-cells measured in blood or tumour samples from patients treated with metronomic cyclophosphamide compared to patients not receiving cyclophosphamide

CONTACTS AND LOCATIONS:
Overall Officials: Freddie Hamdy, Study Chair — Oxford University Hospitals NHS Trust
Locations (2):
- United Kingdom (2):
  - University of Oxford, Oxford
  - Royal Hallamshire Hospital, Sheffield

REFERENCES:
- [Derived] Cappuccini F, Bryant R, Pollock E, Carter L, Verrill C, Hollidge J, Poulton I, Baker M, Mitton C, Baines A, Meier A, Schmidt G, Harrop R, Protheroe A, MacPherson R, Kennish S, Morgan S, Vigano S, Romero PJ, Evans T, Catto J, Hamdy F, Hill AVS, Redchenko I. Safety and immunogenicity of novel 5T4 viral vectored vaccination regimens in early stage prostate cancer: a phase I clinical trial. J Immunother Cancer. 2020 Jun;8(1):e000928. doi: 10.1136/jitc-2020-000928. PMID 32591433